CLINICAL TRIAL: NCT01589484
Title: Impact of Renal Anatomy on Shock Wave Lithotripsy Outcomes for Lower Pole Kidney Stones: Results From a Prospective Multifactorial Analysis
Brief Title: Impact of Renal Anatomy on Shock Wave Lithotripsy Outcomes for Lower Pole Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabio Cesar Miranda Torricelli, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00795812.8.0000.0068
Record Dates: First submitted 2012-04-29; First posted 2012-05-02 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Urolithiasis; Urinary Lithiasis; Kidney Calculi
Keywords: Tomography; Urinary Lithiasis; Kidney Calculi
MeSH Terms: conditions — Urolithiasis; Kidney Calculi | interventions — Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shockwave lithotripsy (SWL) (Experimental): All patients will be submitted to a noncontrast computed tomography before to shockwave lithotripsy (SWL). Patients will be submitted to SWL under the following conditions: outpatient, general anesthesia, 3000 impulses, rate of 90/min, discharged from hospital in the same day with alpha-blocker (doxazosin) during 30 days.
  Interventions: Device: SWL - Compact Delta Dornier Med Tech

INTERVENTIONS:
Device: SWL - Compact Delta Dornier Med Tech — All patients will be submitted to a noncontrast computed tomography before to SWL. Patients will be submitted to SWL under the following conditions: outpatient, general anesthesia, 3000 impulses, rate of 90/min, discharged from hospital in the same day with alpha-blocker (doxazosin) during 30 days.
  Other Names: Extracorporeal shockwave lithotripsy; Compact Delta Dornier Med Tech; Nephrolithotripsy

SUMMARY:
Kidney stone disease affects almost 10% of overall population, often requiring a surgical intervention. Currently, shock wave lithotripsy is considered a first-line treatment option for patients suffering from symptomatic kidney stones smaller than 2.0 cm, providing reasonable stone-free rate. Actually, the outcomes from SWL vary largely due to several factors including stone burden, stone density, stone-skin distance (SSD), and patient's body habitus. Furthermore, the imaging exam modality (i.e. ultrasound versus computed tomography scan) performed to assess the presence of residual fragments also impacts on SWL outcome analysis.

We aim to perform a well-controlled prospective evaluation of all variables that may impact on fragmentation and clearance of lower pole calculi after SWL. These variables are assessed exclusively by a noncontrast computed tomography scan (NCCT), eliminating the necessity of an intravenous urography to study renal collecting system anatomy; an imaging exam that is not routinely performed anymore for kidney stone patients.

DETAILED DESCRIPTION:
Variables in study:

* Age, gender, body mass index (BMI), and waist abdominal circumference
* Noncontrast computed tomography scan (NCCT): stone density (average of 3 measurements), stone size, stone area, skin to stone distance (average of 3 measurements: zero, 45o and 90o), and collecting system anatomy: infundibular length, width, and height, and infundibulopelvic angle

Study design:

All patients will be submitted to a noncontrast computed tomography scan before to SWL. A radiologist with expertise in urolithiasis will evaluate all exams.

Patients will be submitted to SWL under the following conditions: outpatient, general anesthesia, 3000 impulses, rate of 90/min, discharged from hospital in the same day with alpha-blocker (doxazosin) during 30 days.

Patients will be followed up as follow:

* One week after SWL: medical visit To evaluate complications such as pain, dysuria, hematuria, steinstrasse, visit to the emergency department.
* 12 weeks after SWL: new NCCT scan To evaluate kidney stones fragmentation and clearance.

Univariate (Student's T test) and multivariate analysis (multiple logistic regression) will be done to assess the impact of patient's corporal habitus (BMI and abdominal waist circumference), stone characteristics (size, area, density and SSD), and renal collecting system anatomy (infundibular length, width and height, and infundibulopelvic angle) on SWL outcomes (fragmentation and stone-free rates).

ELIGIBILITY:
Inclusion Criteria:

> 17 year-old. Symptomatic single stone of 5 to 20mm located in the lower pole of the kidney. Informed consent signed.

Exclusion Criteria:

Patients with congenital kidney abnormalities (i.e. horseshoes kidney, pelvic kidney, ectopic kidney), patients with ureteral stent (i.e. Double J stent) in the ipsilateral kidney of the stone in study, patients with chronic kidney disease (glomerular filtration rate <60 mL/minute/1.73m2 measured by the equation "Modification of Diet in Renal Disease"), and patients with absolute contraindication to SWL (i.e. coagulopathy, pregnancy, urinary tract infection, or abdominal aneurysm >4.0cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio CM Torricelli, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Shockwave Lithotripsy (SWL): All patients were submitted to a noncontrast computed tomography before to shockwave lithotripsy (SWL). Patients were submitted to SWL under the following conditions: outpatient, general anesthesia, 3000 impulses, rate of 90/min, discharged from hospital in the same day with alpha-blocker (doxazosin) during 30 days.
Period: Overall Study
Arm/Group | Shockwave Lithotripsy (SWL)
Started | 104
Completed | 100
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Shockwave Lithotripsy (SWL): One hundred patients fulfilled the inclusion and exclusion criteria and were enrolled in this study. Mean age and BMI were 47.1 years and 28.0 Kg/m2, respectively. Half of patients had their stone localized in the right kidney. Mean stone size was 9.1mm and mean stone density was 795 HU.
Arm/Group | Shockwave Lithotripsy (SWL)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50
Region of Enrollment [Number; unit: participants]
  Brazil | 100
BMI [Mean (Standard Deviation); unit: Kg/m2] | 28.0 (4.7)
Waist abdominal circumference [Mean (Standard Deviation); unit: cm] | 94.1 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Stone Clearance
Description: After 12 weeks, all patients will be submitted to a new NCCT scan to evaluate stone fragmentation and stone clearance.
Time Frame: 12 weeks after SWL
Population: Fragmentation
Measure: Number; unit: participants
Groups:
- Primary Endoint: Shock wave lithotripsy outcome
Arm/Group | Primary Endoint
Number analyzed (Participants) | 100
participants | 76

2. Secondary Outcome: SWL Complications
Description: Secondary endpoint will be SWL complications (i.e. pain, hematuria, urinary tract infection, Steinstrasse)
Time Frame: 12 weeks after SWL
Measure: Number; unit: participants
Groups:
- SWL Complications: Shock wave lithotripsy complications
Arm/Group | SWL Complications
Number analyzed (Participants) | 100
participants | 7

ADVERSE EVENTS:
Arm/Group | Shockwave Lithotripsy (SWL)
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No